CLINICAL TRIAL: NCT02367417
Title: Prospective Clinical 5-year Follow-up of the LINK® Endo-Model® SL® Rotational and Hinge Knee Prosthesis
Brief Title: Prospective Clinical 5-year Follow-up of the LINK® Endo-Model® SL®
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Waldemar Link GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: RP02
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Bone Necrosis; Arthritis/Arthrosis; Failure of Prosthetic Joint Implant
Keywords: Revision; Knee Joint; PMCF; Endo-Modell SL
MeSH Terms: conditions — Osteonecrosis; Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect outcome information on patients requiring Total Knee Replacement (TKR) in primary or revision cases and therefore receiving the LINK® Endo-Model® SL® under routine conditions.

DETAILED DESCRIPTION:
Post Market Clinical Follow-ups (PMCF) through observational investigations are an important tool to detect infrequent complications or problems, events specific to defined patient populations and long term performance issues under routine condition. Against this background a prospective multi-center study with the LINK® Endo-Model® SL® will be conducted.

ELIGIBILITY:
Inclusion criteria

* Implantation of the LINK® Endo-Model® SL®.
* Between 18 and 78 years of age.
* Patient has signed the Informed Consent. The indications and contraindications for the implantation of the LINK® Endo-Model® SL® listed in the product catalogue and chapter 2.5 and 2.6 [of the protocol] are applicable and have to be considered / fulfilled

Exclusion criteria

* Body Mass Index (BMI) > 40 kg/m2
* Poor general state of health with a foreseeable life expectancy of less than 5 years
* Knee replacement on the contralateral side within the last year and with a KSS fuctional score < 70 points
* Comorbidities and known medical circumstances which forseeable affect the clinical functional results after implantation (e.g. neurological or musculoskeletal impairments)
* Revision in floride septic environment
* Female patient who is pregnant
* Prisoner
* Patient who, as judged by the surgeon, is mentally incompetent or is unlikely to be compliant with the prescribed postoperative routine and follow-up evaluation schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects enrolled in the PMCF in compliance with the inclusion/exclusion criteria who signed the Informed Consent Form and received the Endo-Model SL® prosthesis, will be included in the primary and secondary endpoint analysis.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
KOOS | 1 yr, 3 yrs and 5 yrs
  Knee Injury and Osteoarthritis Outcome Score

SECONDARY OUTCOMES:
Complications | At each Follow-up, up to 5 years
  Rate of implant related, surgery related and systemic complications
Rate of subsequent surgical interventions | At each Follow-up, up to 5 years
  Different surgical interventions
KSS | at 3 months, 1 year and 5 years
  Knee Society Score to assess knee pain and functional knee capacity
Prosthetic Survival Rate | up to 5 years
  Survival of the Prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lohmann, Prof. Dr., Principal Investigator — Medizinische Fakultät Orthopädische Universitätsklinik (KORT), Magdeburg
Locations (3):
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Medizinische Fakultät Orthopädische Universitätsklinik (KORT), Magdeburg, Saxony-Anhalt
  - Evangelisches Waldkrankenhaus Spandau, Berlin

IPD SHARING:
Plan to Share IPD: Undecided